CLINICAL TRIAL: NCT00731159
Title: Sperm Capacitation Assay as a Tool to Predict Sperm Potential to Fertilize in IVF Treatment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Prof A Raziel, Assaf Harofeh MC
Other Study IDs: 54/08
Record Dates: First submitted 2008-08-07; First posted 2008-08-08 (Estimated); Last update posted 2008-08-08 (Estimated); Status verified 2008-07

CONDITIONS: Sperm Capacitation
MeSH Terms: interventions — Sperm Capacitation; Biological Products

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: Sperm capacitation:
  Sperm capacitation is measured in a sample of the same ejaculated sperm unit given for fertilizing human oocytes in an IVF treatment cycle
  Interventions: Biological: sperm capacitation; Other: biologic; Other: sperm capacitation

INTERVENTIONS:
Biological: sperm capacitation — sperm capacitation measured at Bar Ilan University
Other: biologic — sperm synthesis of G-actine to F-actine
  Other Names: sperm capacitation
Other: sperm capacitation — sperm synthesis of G-actine to F-actine
  Other Names: sperm synthesis of G-actine to F-actine

SUMMARY:
Our aim is to evaluate the potential of a new laboratory method that measure sperm capacitation to predict fertilization of oocytes in patients that undergo IVF treatments

DETAILED DESCRIPTION:
Capacitation is a physiologic process in which the sperm acquire the potential to fertilize oocytes. Capacitation can be measured, but the available technics are expensive, inaccurate and complex. A new method to evaluate sperm capacitation was developed in Bar Ilan University, Israel. We intend to measure the capacitation of semen that is used for fertilizing human oocytes in patients treated at the IVF unit at Assaf Harofeh Medical Center.By this, to evaluate the potential of the new method to predict human oocyte fertilization.If the method will be found valuable, it will enable to develop new drugs/methods that may improve sperm capacitation and by this to improve oocyte fertilization leading to more embryos, pregnancies and deliveries.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring IVF within the "routine" work of an IVF Unit
* normo-responding woman
* non ICSI cycles

Exclusion Criteria:

* Patients undergoing ICSI only cycle
* Low responders-less than 8 oocytes
* Male patients with low semen volume

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients requiring IVF within the "routine" work of an IVF Unit
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2008-07; Primary Completion 2009-01 (Estimated); Study Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
Fertilization rate of human oocytes in thr "routine" IVF Laboratory work | One year

CONTACTS AND LOCATIONS:
Locations (1):
- Assaf Harofeh MC, Beer Yaacov, Zerifin, Israel